CLINICAL TRIAL: NCT07295210
Title: Boric Acid Versus 10% Povidone Iodine Solution in Treatment of Otomycosis: a Randomized Clinical Trial
Brief Title: Boric Acid Versus 10% Povidone Iodine Solution in Treatment of Otomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.24.12.3007
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis | interventions — boric acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boric acid group (Active Comparator)
  Interventions: Drug: Boric acid
- Povidone iodine group (Active Comparator)
  Interventions: Drug: Povidone iodine 10%

INTERVENTIONS:
Drug: Boric acid — Boric acid is topically applied to the external auditory canal for treatment of otomycosis
  Arms: Boric acid group
Drug: Povidone iodine 10% — 10% povidone iodine solution is topically applied to the external auditory canal for the treatment of otomycosis
  Arms: Povidone iodine group

SUMMARY:
This study compares two topical agents for the treatment of fungal infection of the external auditory canal: boric acid and a 10% povidone-iodine solution

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients with otomycosis, recruited from the outpatient clinic during the study duration

Exclusion Criteria:

* tympanic membrane perforation
* previous ear surgery
* significant medical co-morbidities such as poorly controlled diabetes or immunocompromised patients
* patient refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
objective clinical response | Days 7, 14, and 28 after treatment
  clinical response is assessed by ear examination by presence or absence of fungal hyphae inside the external auditory canal
Microbiological response | day 28 after treatment
  Microbiological response is evaluated by obtaining cultures from the external auditory canal searching for fungal growth

SECONDARY OUTCOMES:
subjective pain response | days 7, 14, and 28 after treatment
  pain is evaluated on a visual analogue scale from 0 to 10
subjective itching response | days 7, 14, and 28 after treatment
  itching is evaluated on a visual analogue scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Philip A, Thomas R, Job A, Sundaresan VR, Anandan S, Albert RR. Effectiveness of 7.5 percent povidone iodine in comparison to 1 percent clotrimazole with lignocaine in the treatment of otomycosis. ISRN Otolaryngol. 2013 Jul 25;2013:239730. doi: 10.1155/2013/239730. eCollection 2013. PMID 23984100
- [Result] Mofatteh MR, Naseripour Yazdi Z, Yousefi M, Namaei MH. Comparison of the recovery rate of otomycosis using betadine and clotrimazole topical treatment. Braz J Otorhinolaryngol. 2018 Jul-Aug;84(4):404-409. doi: 10.1016/j.bjorl.2017.04.004. Epub 2017 May 6. PMID 28549873
- [Result] del Palacio A, Cuetara MS, Lopez-Suso MJ, Amor E, Garau M. Randomized prospective comparative study: short-term treatment with ciclopiroxolamine (cream and solution) versus boric acid in the treatment of otomycosis. Mycoses. 2002 Oct;45(8):317-28. doi: 10.1046/j.1439-0507.2002.00737.x. PMID 12572722